CLINICAL TRIAL: NCT03973671
Title: Flemish Prospective Clinical and Pathological Database for Urothelial Cancer
Brief Title: Prospective Sample Collection for Cancer of Bladder
Acronym: ProCaB
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S55725
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Risk stratification; Recurrence; Progression; Non-muscle-invasive bladder cancer; Muscle-invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence; Disease Progression; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh-frozen urine, whole blood and bladder cancer tissue (from which DNA/RNA will be extracted in the future).
  These biosamples will be stored at -80°C at the BioBank UZ Leuven.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UC patients: Patients diagnosed with primary or recurrent non-muscle-invasive bladder (NMIBC) cancer.
  No experimental intervention will be administered. NMIBC patients will be diagnosed, treated and followed up according to guidelines-based institutional routines.
  The clinical (demographic, operative and follow-up) and pathological data of the patients will be collected in a complete anonymous way.

SUMMARY:
The goal of the Flemish Databank for Urothelial Cancer is to collect clinical and pathological data of patients treated for urothelial cancer (UC).

DETAILED DESCRIPTION:
The goal of this study is to enable the prospective collection of demographic, clinical, pathological and follow-up data of UC patients after signing informed consent. The specific usage of these prospectively collected clinical data will be described in future trials.

Templates for data collection, which also include clinical outcome parameters and quality indicators, were developed in InfoPath™ as an electronic case report form (eCRF) and were implemented within our hospital's electronic patient file system (called Klinisch Werkstation (KWS), which runs in different Flemish hospitals). These eCRFs have been developed based on the recommendations of the European Association of Urology (EAU) guidelines and the Canadian Urological Association (CUA) white paper. Three separate eCRFs were developed for the management of non-muscle-invasive bladder cancer (NMIBC) patients: surgery report, bladder instillation form, and multidisciplinary team (MDT) form. With the scientific output parameters and quality indicators based on the current knowledge, patient flow-charts for the diagnosis of bladder cancer, and management of low-, intermediate- and high-risk NMIBCs have been developed.

This databank will be first used to externally validate the European Organization for Research and Treatment of Cancer (EORTC) and the Club Urologico Español de Tratamiento Oncologico (CUETO) nomograms for recurrence and progression in patients with NMIBC who have been treated according to the state of the art and prospectively followed up. In-depth analysis of the data generated in this registry will give us the opportunity to define improvements in patient follow-up protocol. Moreover, based on this dataset, we aim to develop a risk calculator for disease recurrence and progression, which will be readily available for Flemish hospitals to use.

ELIGIBILITY:
Inclusion Criteria:

* who are aged between 18-90,
* who are of male or female sex,
* who give their informed consent to collect their clinical and pathological data,
* who are planned to undergo TURBT for BC,
* who are planned to undergo (salvage) radical cystectomy with or without an extended pelvic lymph node dissection,
* who are planned to undergo tumor biopsy (from primary or metastatic tumor),
* who are planned to undergo radical nephroureterectomy ± partial cystectomy or segmental ureterectomy, with or without a lymph node dissection,
* who are planned to undergo endoscopic tumor biopsy or resection,
* from whom metastases will be surgically removed.

Exclusion Criteria:

* patients who do not give their informed consent to collect their clinical and pathological data,
* patients who withdraw their informed consent to use their clinical and pathological data,
* patients who refuse the planned treatment,
* women who are pregnant or have suspicion of pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at University Hospitals Leuven for urothelial cancer that fit the aforementioned inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Progression to MIBC | 10 years
  Histopathologically proven muscle-invasive bladder cancer (at least T2 disease) in pathological evaluation of the TURBT specimen

SECONDARY OUTCOMES:
Recurrence of NMIBC | 5 years
  Clinically (cystoscopically and/or radiologically) proven re-occurence of non-muscle-invasive bladder cancer (Tis, Ta or T1 disease)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joniau, MD, PhD, Principal Investigator — Assistant Professor; Frank Van Der Aa, MD, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No